CLINICAL TRIAL: NCT01995942
Title: Molecular, Pathologic and MRI Investigation of the Prognostic and Redictive Importance of Extramural Venous Invasion in Rectal Cancer
Brief Title: Molecular, Pathologic and MRI Investigation of the Prognostic and Redictive Importance of Extramural Venous Invasion in Rectal Cancer (MARVEL) Trial
Acronym: MARVEL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Pelican Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CCR3873
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Adenocarcinoma; Rectal Diseases; Colorectal Neoplasms; Adenocarcinoma, Mucinous; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Cystic, Mucinous, and Serous; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases
Keywords: Rectal Cancer; EMVI; Extramural Venous Invasion; Microarray; Biomarker; mrEMVI; Tumour Regression Grade; Cancer; Circumferential Resection Margin; CRM; MRI; Radiology; Surgery; Pathology
MeSH Terms: conditions — Adenocarcinoma; Rectal Diseases; Colorectal Neoplasms; Adenocarcinoma, Mucinous; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Cystic, Mucinous, and Serous; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Histopathology samples taken after rectal tumour removal surgery will be analysed using micrarray techniques. The pathological tissue microarrays (TMAs) will be generated using the Alphelys Tissue Arrayer Minicore®3 system. Markers that will be evaluated will be initially directed at epithelial to mesenchymal (EMT) transition pathways, as our preliminary studies suggest that this phylogenetically conserved molecular program has important roles in tumour dissemination and resistance to conventional chemotherapy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Patients with mrEMVI positive rectal cancer
- Group 2: Patients with mrEMVI negative rectal cancer

SUMMARY:
Extramural venous invasion (EMVI) is the spread of microscopic tumour cells into the veins around the tumour. Rectal cancer treatment has improved greatly over recent years. However, it is important for us to learn as much about the tumours as possible in order to develop newer therapies. Current treatments may benefit from new genetic information relating to the cancer. We hope to identify genetic differences in certain types of rectal cancer which will allow future treatments.

DETAILED DESCRIPTION:
Neoadjuvant chemoradiotherapy (CRT) is widely accepted as beneficial to selected patients in terms of decreased risk of local recurrence and overall survival. Current management of rectal cancer involves risk stratification through pre-operative staging leading to formulation of treatment strategy. Very little is known about the long-term outcomes and response to CRT on MRI detected extramural venous invasion (mrEMVI). Although mrEMVI is accepted as a marker of poor prognosis, whether it has a predictive value and should be specifically treated is not known.

Molecular and genetic profiling provides us with an opportunity to understand the underlying mechanisms which govern clinical behaviour in rectal cancer. Using high-throughput technology such as tissue microarray analysis allows large-scale analysis of specimens in a relatively short amount of time. It offers the ability to compare the molecular profiles of different subtypes of rectal cancer such as mrEMVI-positive and -negative tumours and whether any changes are observed following CRT. This can then be correlated with clinical behaviour over the medium and long-term with regards to local recurrence, distant metastases and overall survival.

This study will identify important differences between key rectal cancer tumour subtypes. Identification of reliable pathological markers of EMVI pathways (from both the primary tumour sample, but more importantly from the pre-operative biopsies) has real potential for taking us a step closer to more personalised management of rectal cancer by establishing prognostic biomarkers reflective of disease type, but also through the underlying biology that may be highlighted (with its promise of therapeutic translation).

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced primary rectal cancer (requiring pre-operative treatment); diagnosed on tissue biopsy
2. Adult patients - over 18 years
3. Able to undergo curative (TME) surgery
4. Able to undergo MRI and CT with relevant contrast agent
5. Able to undergo LCRT

Exclusion Criteria

1. Metastatic disease at presentation
2. Emergency diagnosis/treatment
3. Unable to undergo staging (MRI and CT) or treatment procedures (LCRT/surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged over 18 years of age presenting with adenocarcinoma of the rectum. This will be diagnosed on colonoscopy and/or biopsy and MRI, and treatment strategy will include pre-operative CRT followed by surgery.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2013-06-07 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2022-02-02 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be time to relapse pertaining to the primary objective of relapse rate at 1 year and 3 years. | 3 years

SECONDARY OUTCOMES:
Response rates (in terms of mrTstage, mrN stage, involvement of CRM (circumferential resection margin) and mrTRG (tumour regression grade)) in addition to recurrence rates at 1 year and 3 years. | 3 years
Measurement of the change in mrEMVI from pre to post pre-operative therapy, will be based on a new proposed EMVI-TRG classification (EMVI TRG 1-5). | 5 months
  mrEMVI Regression Grade Scoring Table: Grade 5 - No response (intermediate signal intensity, same appearances as original tumour) Grade 4 - Slight response (little areas of fibrosis or mucin but mostly tumour) Grade 3 - Moderate response (>50% fibrosis or mucin, and visible intermediate signal) Grade 2 - Good response (dense fibrosis; no obvious residual tumour, signifying minimal residual disease or no tumour) Grade 1 - Radiological complete response (rCR) (linear/crescentic 1-2mm scar in mucosa or submucosa only.)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Brown, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (19):
- United Kingdom (19):
  - Peterborough City Hospital, Peterborough, Cambridgeshire
  - Leighton Hospital, Crewe, Cheshire
  - Royal Cornwall Hospital, Truro, Cornwall
  - Derriford Hospital, Plymouth, Devon
  - Poole Hospital, Poole, Dorset
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - North Manchester General Hospital, Crumpsall, Manchester
  - University Hospital of South Manchester, Wythenshawe, Manchester
  - Kings Mill Hospital, Sutton in Ashfield, Nottinghamshire
  - Queen's Hospital, Burton Upon Trent, Burton-on-Trent, Staffordshire
  - Royal Surrey County Hospital, Guildford, Surrey
  - Homerton University Hospital, London, Surrey
  - Croydon University Hospital, Thornton Heath, Surrey
  - University Hospital Coventry, Coventry, West Midlands
  - Salisbury District Hospital, Salisbury, Wiltshire
  - Royal Marsden Hospital, London and Surrey
  - George Eliot Hospital, Nuneaton
  - Alexandra Hospital, Redditch
  - South Warwickshire NHS Foundation Trust (Warwick Hospital), Warwick